CLINICAL TRIAL: NCT02926937
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin as Monotherapy in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Efficacy and Safety of Sotagliflozin Versus Placebo in Patients With Type 2 Diabetes Mellitus Not Currently Treated With Antidiabetic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC14833; 2016-001799-31 (EudraCT Number); U1111-1180-6169 (Other: UTN)
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sotagliflozin 400 mg (Experimental): Following a 2-week run-in period, participants were randomized to Sotagliflozin 400 milligrams (mg) administered as two 200 mg tablets, once daily (QD), before the first meal of the day in the double-blind treatment period for up to 26 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954)
- Sotagliflozin 200 mg (Experimental): Following a 2-week run-in period, participants were randomized to Sotagliflozin 200 mg administered as 1 Sotagliflozin tablet and 1 matching placebo tablet, QD, before the first meal of the day in the double-blind treatment period for up to 26 weeks.
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Placebo
- Placebo (Placebo Comparator): Following a 2-week run-in period, participants were randomized to matching placebo to sotagliflozin administered as 2 tablets, QD, before the first meal of the day in the double-blind treatment period for up to 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet;
  Route of administration: oral
  Arms: Sotagliflozin 200 mg; Sotagliflozin 400 mg
Drug: Placebo — Pharmaceutical form: tablet;
  Route of administration: oral
  Arms: Placebo; Sotagliflozin 200 mg

SUMMARY:
Primary Objective:

To demonstrate the superiority of Sotagliflozin 400 milligrams (mg) versus placebo on hemoglobin A1c (HbA1c) reduction in participants with type 2 diabetes (T2D) who have inadequate glycemic control on diet and exercise.

Secondary Objectives:

* To compare Sotagliflozin 400 mg versus placebo based on:
* Change from baseline in 2-hour postprandial glucose (PPG) following a mixed meal.
* Change from baseline in fasting plasma glucose (FPG).
* Change from baseline in systolic blood pressure (SBP) for participants with baseline SBP ≥130 millimeter per mercury (mmHg).
* Change from baseline in SBP for all participants.
* Change from baseline in body weight.
* Proportion of participants with HbA1c <6.5%, <7.0%.
* To compare Sotagliflozin 200 mg versus placebo based on:
* Change from baseline in HbA1c.
* Change from baseline in 2-hour postprandial glucose (PPG) following a mixed meal.
* Change from baseline in body weight.
* Change from baseline in SBP for all participants.
* To evaluate the safety of Sotagliflozin 400 and 200 mg versus placebo.

DETAILED DESCRIPTION:
Up to 34 weeks, including a Screening Period consisting of a Screening Phase of up to 2 weeks and a 2-week single-blind placebo Run-in Phase, a 26-week double-blind Treatment Period, and a 4-week post-treatment Follow-up visit to collect safety information.

ELIGIBILITY:
Inclusion criteria :

* Participants (male and female) with T2D, who are treated with diet and exercise only during the 12 weeks prior to screening.
* Signed written informed consent.

Exclusion criteria:

* Age <18 years at Screening or < legal age of majority, whichever is greater.
* Type 1 diabetes mellitus.
* Body Mass Index (BMI) ≤20 or >45 kilogram per meter square (kg/m^2) at Screening.
* Hemoglobin A1c (HbA1c) <7% or >10% via central laboratory test at Screening.
* Fasting plasma glucose (FPG) >15 millimole per liter (mmol/L) (270 milligram per deciliter [mg/dL]) measured by the central laboratory at screening (Visit 1) and confirmed by a repeat test (>15 mmol/L [270 mg/dL]) before randomization.
* Women of childbearing potential not willing to use highly effective contraceptive method(s) of birth control during the study treatment period and the follow up period or who are unwilling or unable to be tested for pregnancy during the study.
* Treated with an antidiabetic pharmacological agent within the 12 weeks prior to the Screening Visit.
* Previous use of any types of insulin for >1 month (at any time, except for treatment of gestational diabetes).
* History of gastric surgical procedure including gastric banding within 3 years before the Screening Visit.
* History of diabetic ketoacidosis or nonketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* Mean of 3 separate blood pressure measurements >180 millimeter of mercury (mmHg) (systolic) or >100 mmHg (diastolic).
* History of hypertensive emergency within 12 weeks prior to Screening.
* Participants with severe anemia, severe cardiovascular (including congestive heart failure New York Heart Association [NYHA] IV), respiratory, hepatic, neurological, psychiatric, or active malignant tumor or other major systemic disease or participants with short life expectancy that, according to the Investigator, will preclude their safe participation in this study, or will make implementation of the protocol or interpretation of the study results difficult.
* Aspartate aminotransferase and/or alanine aminotransferase: >3 times the upper limit of the normal laboratory range.
* Total bilirubin: >1.5 times the upper limit of the normal laboratory range (except in case of Gilbert's syndrome).
* Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
* Participants who has taken other investigational drugs or prohibited therapy for this study within 12 weeks or 5 half-lives from screening or randomization, whichever is longer. Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research.
* Pregnant (confirmed by serum pregnancy test at Screening) or breastfeeding women.
* Severe renal disease as defined by estimated glomerular filtration rate (eGFR) of <30 millimeter per minute (mL/min)/1.73 meter square (m^2)² at screening by the 4 variable Modification of Diet in Renal Disease (MDRD) equation.
* Participant is unwilling or unable to perform self-monitoring of blood glucose (SMBG), complete the participants diary, or comply with study visits and other study procedures as required per protocol.
* Lower extremity complications (such as skin ulcers, infection, osteomyelitis and gangrene) identified during the Screening period, and still requiring treatment at Randomization.

The above information is not intended to contain all considerations relevant to a Participant potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (70):
- United States (56):
  - Investigational Site Number 8401049, Tucson, Arizona
  - Investigational Site Number 8401026, Tucson, Arizona
  - Investigational Site Number 8401028, Anaheim, California
  - Investigational Site Number 8401057, Canoga Park, California
  - Investigational Site Number 8401058, Garden Grove, California
  - Investigational Site Number 8401029, Hawaiian Gardens, California
  - Investigational Site Number 8401017, Huntington Park, California
  - Investigational Site Number 8401056, Long Beach, California
  - Investigational Site Number 8401013, Long Beach, California
  - Investigational Site Number 8401063, Los Angeles, California
  - Investigational Site Number 8401011, Los Angeles, California
  - Investigational Site Number 8401022, Montclair, California
  - Investigational Site Number 8401039, Norwalk, California
  - Investigational Site Number 8401035, San Dimas, California
  - Investigational Site Number 8401025, Tustin, California
  - Investigational Site Number 8401015, Van Nuys, California
  - Investigational Site Number 8401031, Denver, Colorado
  - Investigational Site Number 8401060, Northglenn, Colorado
  - Investigational Site Number 8401024, Bradenton, Florida
  - Investigational Site Number 8401040, Clearwater, Florida
  - Investigational Site Number 8401014, Daytona Beach, Florida
  - Investigational Site Number 8401007, Hialeah, Florida
  - Investigational Site Number 8401046, Homestead, Florida
  - Investigational Site Number 8401018, Miami, Florida
  - Investigational Site Number 8401008, Miami, Florida
  - Investigational Site Number 8401053, Orlando, Florida
  - Investigational Site Number 8401062, Palm Harbor, Florida
  - Investigational Site Number 8401061, West Palm Beach, Florida
  - Investigational Site Number 8401033, Atlanta, Georgia
  - Investigational Site Number 8401044, Chicago, Illinois
  - Investigational Site Number 8401052, Newton, Iowa
  - Investigational Site Number 8401016, West Des Moines, Iowa
  - Investigational Site Number 8401034, Wichita, Kansas
  - Investigational Site Number 8401038, Lake Charles, Louisiana
  - Investigational Site Number 8401042, Fayetteville, North Carolina
  - Investigational Site Number 8401012, Greensboro, North Carolina
  - Investigational Site Number 8401048, Akron, Ohio
  - Investigational Site Number 8401003, Marion, Ohio
  - Investigational Site Number 8401020, Corvallis, Oregon
  - Investigational Site Number 8401006, Eugene, Oregon
  - Investigational Site Number 8401041, Levittown, Pennsylvania
  - Investigational Site Number 8401051, Anderson, South Carolina
  - Investigational Site Number 8401002, Greer, South Carolina
  - Investigational Site Number 8401005, Fort Worth, Texas
  - Investigational Site Number 8401019, Houston, Texas
  - Investigational Site Number 8401050, Houston, Texas
  - Investigational Site Number 8401037, Katy, Texas
  - Investigational Site Number 8401043, McAllen, Texas
  - Investigational Site Number 8401059, North Richland Hills, Texas
  - Investigational Site Number 8401004, San Antonio, Texas
  - Investigational Site Number 8401054, San Antonio, Texas
  - Investigational Site Number 8401001, San Antonio, Texas
  - Investigational Site Number 8401055, Schertz, Texas
  - Investigational Site Number 8401023, Sugar Land, Texas
  - Investigational Site Number 8401032, Chesapeake, Virginia
  - Investigational Site Number 8401010, Suffolk, Virginia
- Canada (4):
  - Investigational Site Number 1241002, Sherbrooke
  - Investigational Site Number 1241005, Toronto
  - Investigational Site Number 1241001, Toronto
  - Investigational Site Number 1241006, Vancouver
- Mexico (10):
  - Investigational Site Number 4841006, Aguascalientes
  - Investigational Site Number 4841010, Aguascalientes
  - Investigational Site Number 4841003, Cd. México, México
  - Investigational Site Number 4841004, Chihuahua City
  - Investigational Site Number 4841001, Culiacán
  - Investigational Site Number 4841005, Durango, Durango
  - Investigational Site Number 4841009, Guadalajara
  - Investigational Site Number 4841007, México
  - Investigational Site Number 4841008, Monterrey
  - Investigational Site Number 4841002, Monterrey, Nuevo León

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 70 investigative sites in the United States, Canada, Mexico, from 11 November 2016 to 17 May 2019.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled in 1 of 3 treatment groups: Placebo, Sotagliflozin 400 milligrams (mg) or Sotagliflozin 200 mg.
Groups:
- Placebo: Following a 2-week run-in period, participants were randomized to matching placebo to sotagliflozin administered as 2 tablets, once daily (QD), before the first meal of the day in the double-blind treatment period for up to 26 weeks.
- Sotagliflozin 400 mg: Following a 2-week run-in period, participants were randomized to Sotagliflozin 400 mg administered as two 200 mg tablets, QD, before the first meal of the day in the double-blind treatment period for up to 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg
Started | 150 | 142 | 107
Completed | 131 | 127 | 96
Not Completed | 19 | 15 | 11
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Poor Compliance to Protocol | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 5 | 0
Not completed — At the Participant's own Request | 11 | 5 | 8
Not completed — Reason not Specified | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The randomized population included any participant who had been allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg | Total
Number analyzed (Participants) | 150 | 142 | 107 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.2) | 54.7 (11.2) | 52.3 (11.4) | 54.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 68 | 53 | 193
  Male | 78 | 74 | 54 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 85 | 69 | 253
  Not Hispanic or Latino | 51 | 57 | 36 | 144
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 3 | 3 | 18
  Asian | 9 | 4 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 18 | 12 | 47
  White | 112 | 117 | 77 | 306
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 13 | 7 | 31
  United States | 96 | 100 | 63 | 259
  Mexico | 43 | 29 | 37 | 109
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.11 (0.88) | 8.14 (0.92) | 8.00 (0.81) | 8.09 (0.87)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 127.27 (13.08) | 128.70 (4.80) | 128.08 (13.08) | 128.00 (13.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Description: An analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Participants in the Intent-to-treat (ITT) population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
percentage of HbA1c | -0.34 (0.120) | -1.03 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares (LS) Mean = -0.69, 95% CI 2-sided [-0.975 to -0.415]

2. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose (PPG) Following a Mixed Meal at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
millimole per liter (mmol/L) | -0.591 (0.1943) | -1.156 (0.1964)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, country, treatment-by-country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.0141, ANCOVA; Difference in LS Mean = -0.565, 95% CI 2-sided [-1.0166 to -0.1140]

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose (PPG) Following a Mixed Meal at Week 26 (Sotagliflozin 200 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 200 mg and Placebo under Protocol Amendment 1. Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 110 | 107
mmol/L | -0.500 (0.2443) | -0.847 (0.2477)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups under Amendment 1 randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, country, treatment-by-country as fixed effects, and baseline HbA1c as a covariate; Test type: Superiority; p = 0.2081, ANCOVA; Difference in LS Mean = -0.346, 95% CI 2-sided [-0.8853 to 0.1928]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1.Missing data are imputed using washout imputation method under the missing not at random framework.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
mmol/L | -0.201 (0.2739) | -1.756 (0.2719)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥ 130mmHg) at screening, and country as fixed effects, and baseline fasting plasma glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = -1.556, 95% CI 2-sided [-2.1876 to -0.9234]

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 12 in Participants With Baseline SBP ≥130 Millimeter of Mercury (mmHg) (Sotagliflozin 400 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: Analysis was performed on participants in the ITT population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1 with Baseline SBP ≥130 mmHg. Missing data are imputed using washout imputation method under the missing not at random framework. This Outcome Measure was pre-specified in the protocol to be assessed in the Placebo and Sotagliflozin 400 mg arms.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 55 | 48
mmHg | -4.45 (2.419) | -7.96 (2.282)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 12 is analyzed using analysis ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.1680, ANCOVA; Difference in LS Mean = -3.50, 95% CI 2-sided [-8.478 to 1.476]

6. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants (Sotagliflozin 400 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
mmHg | -0.57 (1.088) | -1.35 (1.116)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 12 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline SBP as a covariate; Test type: Superiority; p = 0.5467, ANCOVA; Difference in LS Mean = -0.78, 95% CI 2-sided [-3.311 to 1.753]

7. Secondary Outcome: Change From Baseline in SBP at Week 12 for All Participants (Sotagliflozin 200 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 110 | 107
mmHg | -1.62 (1.215) | -4.82 (1.211)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0193, ANCOVA; Difference in LS Mean = -3.19, 95% CI 2-sided [-5.869 to -0.518]

8. Secondary Outcome: Change From Baseline in Body Weight at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram (Kg)
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
kilogram (Kg) | -0.79 (0.373) | -2.33 (0.379)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130 mmHg) at screening, and country as fixed effects, and baseline weight as a covariate; Test type: Superiority; p = 0.0005, ANCOVA; Difference in LS Mean = -1.54, 95% CI 2-sided [-2.404 to -0.676]

9. Secondary Outcome: Change From Baseline in Body Weight at Week 26 (Sotagliflozin 200 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 110 | 107
kg | -0.52 (0.509) | -1.69 (0.518)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; The change from baseline to Week 26 is analyzed using ANCOVA model with treatment groups, randomization strata of HbA1c (≤8.0, >8.0%) at screening, randomization strata of mean SBP (<130, ≥130mmHg) at screening, and country as fixed effects, and baseline weight as a covariate; Test type: Superiority; p = 0.0406, ANCOVA; Difference in LS Mean = -1.17, 95% CI 2-sided [-2.281 to -0.050]

10. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Time Frame: Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1. This Outcome Measure was pre-specified in the protocol to be assessed in the Placebo and Sotagliflozin 400 mg arms.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
percentage of participants | 10.7 | 23.2
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; Percentage difference between treatment groups from each stratum (randomization strata of HbA1c (<=8.0, >8.0%) at screening, randomization strata of mean SBP (<130, >=130 mmHg) at screening) using Cochran-Mantel-Haenszel weights; Test type: Superiority; p = 0.0037, Cochran-Mantel-Haenszel; Percentage Difference = 12.6, 95% CI 2-sided [4.18 to 21.02]

11. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 26 (Sotagliflozin 400 mg Versus Placebo)
Time Frame: Week 26
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
percentage of participants | 28.0 | 47.2
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Percentage Difference = 19.2, 95% CI 2-sided [8.39 to 30.00]

12. Secondary Outcome: Change From Baseline in HbA1c at Week 26 (Sotagliflozin 200 mg Versus Placebo)
Description: An ANCOVA model was used for the analysis.
Time Frame: Baseline to Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 110 | 107
percentage of HbA1c | -0.26 (0.143) | -0.93 (0.148)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS Mean = -0.67, 95% CI 2-sided [-0.989 to -0.354]

13. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events (Sotagliflozin 400 mg Versus Placebo)
Description: Percentage of participants with hypoglycemic events are reported for the following 3 categories: Any hypoglycemia (as reported in the Electronic Case Report Form); Documented symptomatic hypoglycemia [typical symptoms of hypoglycemia (increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, and/or coma) and plasma glucose ≤70 mg/dL (3.9 mmol/L)]; Severe [an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions] or documented symptomatic hypoglycemia [typical symptoms of hypoglycemia and plasma glucose ≤70 mg/dL]. Participants may be reported in more than one category.
Time Frame: Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 400 mg and Placebo under original Protocol and Protocol Amendment 1.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 400 mg
Number analyzed (Participants) | 150 | 142
percentage of participants
  Any hypoglycemia | 2.7 | 2.1
  Documented symptomatic hypoglycemia | 1.3 | 0.7
  Severe or documented symptomatic hypoglycemia | 1.3 | 0.7

14. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemic Events (Sotagliflozin 200 mg Versus Placebo)
Description: as for outcome 13
Time Frame: Week 26
Population: Participants in the ITT population who were randomized to Sotagliflozin 200 mg and Placebo under Protocol Amendment 1.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg
Number analyzed (Participants) | 110 | 107
percentage of participants
  Any hypoglycemia | 2.7 | 1.9
  Documented symptomatic hypoglycemia | 0.9 | 0.9
  Severe or documented symptomatic hypoglycemia | 0.9 | 0.9

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose of study drug (up to 26 weeks) + 4 weeks
Description: Safety population included all randomized participants who had received at least one dose of double-blind investigational medicinal product (IMP).
Arm/Group | Placebo | Sotagliflozin 400 mg | Sotagliflozin 200 mg
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/142 | 0/107
Serious Adverse Events (participants affected / at risk) | 3/150 | 3/142 | 2/107
Other Adverse Events (participants affected / at risk) | 20/150 | 17/142 | 14/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | Sotagliflozin 400 mg (N=142) | Sotagliflozin 200 mg (N=107)
Retinal detachment (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | Sotagliflozin 400 mg (N=142) | Sotagliflozin 200 mg (N=107)
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 5
Urinary tract infection (Infections and infestations) | 7 | 8 | 3
Headache (Nervous system disorders) | 9 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02926937/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT02926937/SAP_001.pdf